CLINICAL TRIAL: NCT04221386
Title: Melodic Intonation Therapy for Tone Language Speakers
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Coronavirus
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IZZKJ
Record Dates: First submitted 2020-01-03; First posted 2020-01-09 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2019-12

CONDITIONS: Dementia; Speech Therapy
Keywords: Melodic Intonation Therapy; Music; Tone language
MeSH Terms: conditions — Dementia; Communication Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIT group (Experimental): Subjects will receive the developed Melodic Intonation Therapy.
  Interventions: Behavioral: Melodic Intonation Therapy (MIT)
- Control group (No Intervention): Subjects will not receive any intervention.

INTERVENTIONS:
Behavioral: Melodic Intonation Therapy (MIT) — Subjects will receive at least 6 MIT sessions in group of 3-5 subjects. In the sessions, experimenter will sing songs with the subjects. Songs used in the intervention are familiar to elderly and are rewritten and embedded with everyday phrases and vocabularies. The whole intervention will span 3-4 weeks.
  Arms: MIT group

SUMMARY:
One of the traditional therapies for restoring the ability of speech in aphasic patients is Melodic Intonation Therapy (MIT), in which everyday phrases are taught in a singing-like manner. The suggested mechanism for speech recovery is that because of the sharing of brain resources for language and music, the regions normally reserved for singing can be trained to help compensate the speech functions originally subserved by the damaged regions. However, this therapy has primarily been applied to speakers of non-tone languages, in which prosodic features carry a more important role than pitch features in conveying meanings. It remains unknown whether MIT will be equally applicable for speakers of tone languages, in which pitch features likely play a more important role. Another uncertainty concerns whether the efficacy of MIT can be extended to patients with expressive speech impairment due to dementia. This pilot study aims to find out the efficacy of MIT for speech-impaired dementia patients in different verbal tasks. The results of this study will provide preliminary empirical evidence to establish the utility of MIT for Cantonese speakers in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Early to moderate stage dementia patient
* Normal hearing (hearing aid accepted)
* Non-fluent speech (max. score of fluency in Cantonese Aphasia Battery spontaneous speech subtest = 6/10)

Exclusion Criteria:

* Non-native Cantonese speaker
* Illiterate
* Aphasic patients
* Subjects who receive other speech therapy during study

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Aphasia Quotient (AQ) in Cantonese Aphasia Battery | within a week after procedure
  Two subtests of the Cantonese Aphasia Battery (auditory comprehension & spontaneous speech) will be executed. Higher AQ means better performance in the respective areas. The minimum of AQ in each subtest is 0, and the maximum is 20.

SECONDARY OUTCOMES:
Change in latency and accuracy in picture naming task | within a week after procedure
  In the computerized picture naming task, subjects are asked to name the objects they see in 52 pictures, within 5000 ms per picture. Visual stimuli of the task are black and white line-drawings. Responses are all recorded for analysis.
Change in performance of semantic fluency task | within a week after procedure
  In the computerized semantic fluency task, subjects are given 5 categories (e.g. animals) and asked to name as many members of the categories (e.g. cat, dog) as possible. For each category, they have one minute to respond. All the responses are recorded for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: William Shi Yuan Wang, Ph.D., Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Elderly homes, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
All the data collected in screening, pre- and post-assessment will not be shared with other researchers.

REFERENCES:
- [Background] Albert ML, Sparks RW, Helm NA. Melodic intonation therapy for aphasia. Arch Neurol. 1973 Aug;29(2):130-1. doi: 10.1001/archneur.1973.00490260074018. No abstract available. PMID 4717723
- [Background] Sparks R, Helm N, Albert M. Aphasia rehabilitation resulting from melodic intonation therapy. Cortex. 1974 Dec;10(4):303-16. doi: 10.1016/s0010-9452(74)80024-9. No abstract available. PMID 4452250
- [Result] Sarkamo T, Sihvonen AJ. Golden oldies and silver brains: Deficits, preservation, learning, and rehabilitation effects of music in ageing-related neurological disorders. Cortex. 2018 Dec;109:104-123. doi: 10.1016/j.cortex.2018.08.034. Epub 2018 Sep 19. PMID 30312779